CLINICAL TRIAL: NCT06120920
Title: Comparison of Hip Strengthening Exercises and Core Stability Exercises in Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-545-10-2023
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Knee Osteoarthritis
Keywords: Hip Strengthening Exercises; Core Stability Exercises; Routine Knee Strengthening Exercises; Conventional Physical Therapy; Pain Assessment; Range of Motion; Functional Disability; Knee Muscle Strength; Time Up and Go Test
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be unaware of the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physical Therapy and Routine Knee Exercises with Core Stability Exercises. (Active Comparator): Patient will receive Conventional physical therapy include hot pack, Tens and routine knee strengthening exercises with core stability exercises.
  Interventions: Other: Assigned Interventions; Other: Conventional Physical Therapy and Routine Knee Exercises with Hip Strengthening Exercises.
- Conventional Physical Therapy and Routine Knee Exercises with Hip Strengthening Exercises. (Experimental): In this group, patient will receive conventional physical therapy include hot pack, Tens and routine knee exercises with hip strengthening exercises
  Interventions: Other: Assigned Interventions; Other: Conventional Physical Therapy and Routine Knee Exercises with Hip Strengthening Exercises.

INTERVENTIONS:
Other: Assigned Interventions — Conventional physical therapy consists of hot pack application and transcutaneous electric stimulation (TENS) and routine knee strengthening exercises in addition with core stability exercises in three sessions per week for 4 weeks. Core stability exercises include bent knee hollow hold, bridging, supine toe tap and knee strengthening exercises include knee flexion strengthening exercises and knee extension isometric exercises.
  Other Names: Conventional Physical Therapy and Routine Knee Exercises with Core Stability Exercises.
Other: Conventional Physical Therapy and Routine Knee Exercises with Hip Strengthening Exercises. — Conventional physical therapy consists of hot pack application, Tens and routine knee exercise program same as group A and in addition with hip strengthening exercises. Hip strengthening exercises include hip flexion and extension strengthening exercises and hip internal rotation and external rotation and hip adduction and abduction strengthening exercises.C

SUMMARY:
Knee Osteoarthritis is a chronic degenerative joint disease with complex etiology that results in loss of normal joint function due to damage to the articular cartilage. It is characterized by pain, swelling, inflammation and narrowing in articular cartilage. Hip muscle weakness has been observed in persons with knee OA and poor core stability may be one of the other contributing factors that lead to knee OA development as well as its progression. Core stabilization and muscular synergism of the trunk and hip work is an effective way to improve lower limb strength balance and prevent injury. So the lumbopelvic stability is vital to support loads on the knee joint.

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the knee joint results in chronic pain and functional decline among older adults. Osteoarthritis is a degenerative joint disease with complex etiology that results in loss of normal joint function due to narrowing of the articular cartilage. The pathogenesis of knee OA is the result of interaction between mechanical loading, articular cartilage damage, and incomplete repair mechanisms. These changes eventually cause progressive joint degeneration and failure, leading to chronic knee pain and progressive restriction of knee joint mobility. Core muscle endurance deficiency leads to an increase in the loading of the knee, as well as in knee joint contact force during dynamic movement. Hence, poor core stability may be one of the contributing factors that lead to knee OA development as well as its progression. On the other hand hip muscle weakness has been observed in persons with knee OA and to increase the medial compartment loading on the knee joint. This increases the force on the medial compartment of the stance leg, and the disease starts succeeding. Core stabilization and muscular synergism of the trunk and hip work is an effective way to improve lower limb strength balance and prevent injury. Considering the strength deficits in the hip muscles as well as core muscles, a targeted exercise program for knee osteoarthritis include hip muscle strengthening and core strengthening might reduce the medial compartment loading and improve knee symptoms. Core stability and hip strengthening exercise along with Knee Physical therapy and conventional therapy as a mode of treatment in knee OA and it may help clinicians to treat subjects with knee OA at risk of a decline in muscle strength, range of motion, functional disability and pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 40-65
2. Diagnose case of knee OA grade 2, 3.
3. Side of involved leg: right or left.
4. Unilateral knee.
5. Gender both male and female.
6. Pre-diagnostics referred by orthopedics.
7. Able to walk without gait aids.

Exclusion Criteria:

1. Inflammatory arthritis
2. Osteoarthritis of the hips
3. Having had previous knee or hip surgery.
4. Patient who had amputated leg and who don't have any lower extremity disorders.
5. Received intra-articular injection within 6 months.
6. Non-steroidal anti-inflammatory drug or cortisone use over an extended period.
7. Patients who had neurological and muscle problem

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2023-11-21 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Pain Assessment | Pain intensity will be measured at the baseline at the time of recruitment and change in pain intensity will be measured at 3rd and 4th week of interventions
  Pain intensity will be measured using Visual Analogue Scale. It consist of a 100mm line, with to end points, 0 representing no pain and 10 representing pain as bad as it could be possible.
Knee Range of Motion | Knee Range of Motion will be measured as baseline at the time of recruitment and change in range of motion will be measured at 3rd and 4th week of treatment.
  ROM is measured by goniometer.: A normal range of knee joint is 0 degrees of knee extension (a fully straightened knee) and 135 degrees of knee flexion.A half circle long-arm metallic goniometer, ranging from 0 to 180°, with 1° interval marking was used. It had a central fulcrum, a stationary or fixed arm, and a pivoting or moving arm. Both arms were 30 cm long.
Functional Disability | Level of Functional Disability will be recorded as baseline at the time of recruitment and change in functional status will be observed at the 3rd and 4th week of intervention.
  The functional disability assessed by the self-reported questionnaire the Knee injury and Osteoarthritis Outcome Score (KOOS).Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.
Knee Muscle Strength | Knee Muscle Strength will be observed as baseline at the time of recruitment and change in muscle strength will be observed at the 3rd and 4th week of treatment
  Knee Muscle Strength will be observed by Manual Muscle Testing Scale. This method involves testing key muscles from the lower extremities against the examiner's resistance and grading the patient's strength on a 0 to 5 scale accordingly 1.Flicker of movement,2.through full range actively with gravity counterbalanced,3.through full range actively against gravity,4.through full range actively against some resistance,5.Through full range actively against strong resistance.

SECONDARY OUTCOMES:
Timed Up and Go Test (TUG) | Time Up and Go Test will be observed as baseline at the time of recruitment and change in function will be observed at 3rd and 4th week of treatment.
  TUG is used to evaluate function. It assesses the patient's capability to stand from the chair, then walk for three meters, turn, walk back, and sit on the same chair. The TUG is highly responsive and valid to determine alteration in patients with OA of the knee. The minimum clinically important differences (MCID) is reported to be 0.8-1.4s for the TUG in patients with OA of the knee.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Waqar Afzal, PhD, Study Chair — University of Lahore
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Participants data that underlies the results after de-identification.
Supporting Information: Study Protocol
Time Frame: Immediately after publication
Access Criteria: Researchers who provide methodological sound proposal